CLINICAL TRIAL: NCT05626959
Title: A Phase II/III Double-Blind, Randomised and Controlled-to-Open-Label Study Assessing the Efficacy of Full-Spectrum Medicinal Cannabis Plant Extract 0.08% THC (NTI164) on the Severity of Autism Spectrum Disorder in Young People
Brief Title: Evaluating the Efficacy of NTI164 in Young People With Autism Spectrum Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fenix Innovation Group (Industry)
Collaborators: Neurotech International Limited (Industry); Monash Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NTIASD2
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: At the beginning of the study, participants will be randomised into either the active group or placebo group. Both groups will commence a double-blinded baseline dose of either 5mg/kg/day of NTI164 or Placebo that will be increased weekly by 5mg/kg for a period of 4 weeks until the maximum tolerated dose or 20/mg/kg/day is achieved.
  At the end of the 8-week period, both study groups will be unblinded and all participants will begin or continue NTI164 for 8 weeks.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Allocation is concealed utilising central randomisation by computer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NTI164 (Experimental): Full-Spectrum Medicinal Cannabis Plant Extract with less than 0.08% THC (NTI164)
  Randomised Controlled Phase:
  Part A: 5mg/kg, 10mg/kg, 15mg/kg, 20mg/kg (1 week each, total duration = 4 weeks) Part B: 20mg/kg or maximum tolerated dose (total duration = 4 weeks).
  Open-Label Phase 20mg/kg or maximum tolerated dose (total duration = 8 weeks).
  Extension Phase 20mg/kg or maximum tolerated dose (total duration = 36 weeks).
  Interventions: Drug: NTI164
- Placebo (Placebo Comparator): Randomised Controlled Phase:
  Part A: 5mg/kg, 10mg/kg, 15mg/kg, 20mg/kg (1 week each, total duration = 4 weeks) Part B: 20mg/kg or maximum tolerated dose (total duration = 4 weeks).
  Interventions: Drug: NTI164

INTERVENTIONS:
Drug: NTI164 — Oil based. Full-spectrum medicinal cannabis plant extract with less than 0.08% THC.
  Other Names: Full-spectrum medicinal cannabis plant extract 0.08% THC

SUMMARY:
This is an 18 to 54 week study assessing the efficacy of Full-Spectrum Medicinal Cannabis Plant Extract 0.08% THC (NTI164) on the severity of autism spectrum disorder in young people.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of NTI164 in patients with ASD when treated with 20mg/kg/day for 8 - 54 weeks.

The study comprises of an 8-week double-blinded randomised controlled treatment period followed by an 8-week open-label maintenance period followed by a 2-week wash-out period. Participants who wish to continue receiving the study treatment beyond the 16 week period may do so for up to fifty-two weeks (Extension phase).

Efficacy will be measured and monitored by performing participant- and psychologist- led questionnaires specific to measuring changes in the behaviour of patients with ASD.

Safety will be measured and monitored by performing full blood examinations and liver and renal function tests throughout the study.

Additional assessments include microbiome and inflammatory marker assessments.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant is aged 8 years to 17 years (inclusive)
* Participant is at a healthy weight at the discretion of the Principal Investigator.
* Parents or caregivers can give informed consent for participation in the trial with assent from individuals with autism.
* Participants can comply with trial requirements.
* According the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria the participant has a diagnosis of Level 2 or 3 Autism Spectrum Disorder (ASD) confirmed by Autism Diagnostic Observational Schedule (ADOS-2) criteria
* All treatments including medications and therapies for ASD related symptoms must have been stable for 4 weeks before enrolment and for the duration of the trial wherever possible.
* Participants must be able to swallow liquid.
* Consent giver must be able to understand the requirements of the study.

EXCLUSION CRITERIA:

* Current diagnosis of bipolar disorder, psychosis, schizophrenia, schizoaffective disorder, or active major depression
* Has a diagnosis other than ASD that dominates the clinical presentation (e.g., Attention Deficit Hyperactivity Disorder [ADHD])
* Has a degenerative condition
* Changes in anticonvulsive therapy within the last 12 weeks
* Taking omeprazole, lansoprazole, tolbutamide, warfarin, sirolimus, everolimus, temsirolimus, tacrolimus, clobazam, repaglinide, pioglitazone, rosiglitazone, montelukast, bupropion, or efavirenz
* Currently using or has used recreational or medicinal cannabis, cannabinoid-based medications (including Sativex®, or Epidiolex®) within the 12 weeks prior to screening and is unwilling to abstain for the duration of the trial
* Participant has any known or suspected hypersensitivity to cannabinoids or any of the excipients
* Participant has moderately impaired hepatic function at screening, defined as serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2 × upper limit of normal (ULN) or total bilirubin (TBL) > 2 × ULN. This criterion can only be confirmed once the laboratory results are available; participants enrolled into the trial who are later found to meet this criterion must be screen-failed.
* Participant is male and fertile (i.e., after puberty unless permanently sterile by bilateral orchidectomy) unless willing to ensure that they use male contraception (condom) or remain sexually abstinent during the trial and for 12 weeks thereafter.
* Participant is female and with childbearing potential (i.e., following menarche and until becoming postmenopausal for greater than or equal to 12 consecutive months unless permanently sterile by hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) unless willing to ensure that they use a highly effective method of birth control (e.g., hormonal contraception, intrauterine device/hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence) during the trial and for 12 weeks thereafter.
* Female participant who is pregnant (positive pregnancy test), lactating or planning pregnancy during the course of the trial or within 12 weeks thereafter.
* Participant had brain surgery or traumatic brain injury within 1 year of screening.
* Participant has any other significant disease or disorder which, in the opinion of the investigator, may either put the participant, other participants, or site staff at risk because of participation in the trial, may influence the result of the trial, or may affect the participant's ability to take part in the trial.
* Any abnormalities identified following a physical examination of the participant that, in the opinion of the investigator, would jeopardize the safety of the participant if they took part in the trial
* Any history of suicidal behaviour (lifelong) or any suicidal ideation of type 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the last 4 weeks or at screening or randomization
* Participant has donated blood during the past 12 weeks and is unwilling to abstain from donation of blood during the trial.
* Participant has any known or suspected history of alcohol or substance abuse or positive drugs of abuse test at screening (not justified by a known concurrent medication).
* Participant has previously been enrolled into this trial.
* Participant has plans to travel outside their country of residence during the trial, unless the participant has confirmation that the product is permitted in the destination country/state.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2022-11-30 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Global Impression-Severity (CGI-S) | Baseline, Week 8.
  Reflects clinician's impression of severity of illness on a 7-point scale ranging from 1=not at all to 7=among the most extremely ill.

SECONDARY OUTCOMES:
Vineland Adaptive Behaviour Scales, Third Edition | Baseline, Weeks 16, 28, 40 & 52
  Used to measure adaptive functioning across three core domains (Communication, Daily Living Skills, and Socialization), and two optional domains (Motor Skills and Maladaptive Behaviour); items are rated on a 3-point scale (0=never; 1=sometimes; 2=usually or often). The core domains sum to a total Adaptive Behaviour Composite.
Social Responsiveness Scale, 2nd Editions (SRS-2) | Baseline, Weeks 16, 28, 40 & 52
  Five domains are assessed including: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behaviour. Items are scored on a 4-point scale (ranging from 1=not true to 4=almost always true).
Clinical Global Impression Scale - Improvement (CGI-I) | Baseline, Weeks 4, 8, 12, 16, 28, 40 & 52
  This is a 7-point scale measuring symptom change from baseline.
Anxiety, Depression and Mood Scale (ADAMS) | Baseline, Weeks 16, 28, 40 & 52
  28 symptom items that resolve into five subscales labelled: Manic/Hyperactive Behaviour, Depressed Mood, Social Avoidance, General Anxiety, and Compulsive Behaviour. Items are rated on 4-point scale ranging from 0=not a problem to 3=severe problem.
Sleep Disturbance Scale for Children (SDSC) | Baseline, Weeks 4, 8, 12, 16, 28, 40 & 52
  Six subscales including Disorders of Initiating and Maintaining Sleep, Sleep Breathing Disorders, Disorders of Arousal, Sleep Wake Transition Disorders, Disorders of Excessive Somnolence, and Sleep Hyperhydrosis. Items are rated on 5-point scale where 1=never and 5=always (daily). Subscale scores sum to equal a total score
Anxiety Scale for Children - Autism Spectrum Disorder | Baseline, Weeks 4, 8, 12, 16, 28, 40 & 52
  A form developed to detect symptoms of anxiety in youth with ASD. Composed of four subscales (Performance Anxiety, Uncertainty, Anxious Arousal, and Separation Anxiety), items are rated on a 4-point scale (0=never and 3=always). Subscales sum to equal a total score.
Caregiver Global Impression of Change in Attention (CGI-CA) | Baseline, Weeks 4, 8, 12, 16, 28, 40 & 52
  Reflects clinician's impression of change in attention on a 7-point scale ranging from 1=not at all to 7=very severe problem. Provided as Baseline and Post-Baseline questionnaires.
Caregiver Global Impression of Change (CGI-C) Target Behaviour | Baseline, Weeks 4, 8, 12, 16, 28, 40 & 52
  Reflects clinician's impression of change of behaviour on a 7-point scale ranging from 1=not at all to 7=very severe problem. Provided as Baseline and Post-Baseline questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fahey, Prof, Principal Investigator — Head of Paediatric Neurology
Locations (1):
- Monash Children's Hospital, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No